CLINICAL TRIAL: NCT00226096
Title: A Randomised Trial to Establish the Effects of Early Intensive Blood Pressure Lowering on Death and Disability in Patients With Stroke Due to Acute Intracerebral Haemorrhage
Brief Title: Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDA1INTERACT
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: CVA (Cerebrovascular Accident); Cerebral Hemorrhage; Intracranial Hemorrhages
Keywords: Clinical Trial; Blood Pressure; CVA (Cerebrovascular Accident)
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Intracranial Hemorrhages | interventions — Labetalol; Metoprolol; Hydralazine; Nitroglycerin; Phentolamine; Nicardipine; urapidil; esmolol; Clonidine; Enalaprilat; Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Labetalol Hydrochloride
Drug: Metoprolol tartrate
Drug: Hydralazine Hydrochloride
Drug: Glycerol Trinitrate
Drug: Phentolamine mesylate
Drug: Nicardipine
Drug: Urapidil
Drug: Esmolol
Drug: Clonidine
Drug: Enalaprilat
Drug: Nitroprusside

SUMMARY:
The purpose of the study is to determine whether lowering high blood pressure levels after the start of a stroke caused by bleeding in the brain (intracerebral haemorrhage) will reduce the chances of a person dying or surviving with a long term disability. The study will be undertaken in two phases: a vanguard phase in 400 patients, to plan for a main phase in 2000 patients.

DETAILED DESCRIPTION:
Intracerebral haemorrhage (ICH) is one of the most serious subtypes of stroke, affecting approximately 2-3 million people worldwide each year. About one third of people with ICH die early after onset and the majority of survivors are left with major long-term disability. Administration of activated recombinant human Factor VII has been shown to limit haematoma expansion in randomised controlled clinical trials; however, future clinical use of this agent may be limited by a short therapeutic time window, contraindication in patients at risk of thromboembolism and high cost. Currently, no acute medical therapies have been shown to alter outcome in ICH and the role of surgery remains uncertain.

Blood pressure (BP) levels are strongly and positively associated with the incidence of first and recurrent stroke and there is definite evidence that BP lowering reduces stroke risk. Although BP levels are commonly elevated after stroke onset, particularly in ICH, the effects of BP lowering treatment in the acute phase of stroke remain unknown.

The study aims to establish the effectiveness of a management policy of early intensive BP lowering on death & disability in patients with primary ICH compared to current guideline-based management of high BP in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Acute stroke due to spontaneous ICH confirmed by clinical history & CT scan
* At least 2 systolic BP measurements of >/=150mmHg and </=220mmHg, recorded 2 or more minutes apart
* Able to commence randomly assigned BP lowering regimen within 6 hours of stroke onset
* Able to be actively treated and admitted to a monitored facility e.g. HDU/ICU/acute stroke unit

Exclusion Criteria:

* Known definite contraindication to an intensive BP lowering regimen
* Known definite indication for intensive BP lowering regimen as (or more) intensive than the active treatment arm
* Definite evidence that the ICH is secondary to a structural abnormality in the brain
* Previous ischaemic stroke within 30 days
* A very high likelihood that the patient will die within the next 24 hours on the basis of clinical and/or radiological criteria
* Known advanced dementia or significant pre-stroke disability
* Concomitant medical illness that would interfere with outcome assessments and follow up
* Already booked for surgical evacuation of haematoma
* Previous participation in this trial or current participation in another investigational drug trial
* A high likelihood that the patient will not adhere to the study treatment and follow up regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Combination death and dependency, according to a 3-6 scores on the modified Rankin Score. | 3 months

SECONDARY OUTCOMES:
All cause and cause-specific early neurological deterioration during the first 72 hours; haematoma expansion & cerebral oedema at 24 & 72 hours; ; functional disability; cognitive function; quality of life; mortality at 1 and 3 months | 24 and 72 hours, 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, PhD, Principal Investigator — The George Institute; Bruce Neal, PhD, Principal Investigator — The George Institute
Locations (20):
- Australia (15):
  - Concord Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- China (3):
  - Regional Coordinating Centre: Peking University First Hospital, Beijing
  - Hospitals in China, c/o The George Institute China, Beijing
  - Regional Coordinating Centre: Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai Institute of Hypertension, Shanghai Second Medical University, Shanghai
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Result] Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J; INTERACT Investigators. Intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT): a randomised pilot trial. Lancet Neurol. 2008 May;7(5):391-9. doi: 10.1016/S1474-4422(08)70069-3. Epub 2008 Apr 7. PMID 18396107
- [Derived] Wang X, Ren X, Li Q, Ouyang M, Chen C, Delcourt C, Chen X, Wang J, Robinson T, Arima H, Ma L, Hu X, You C, Li G, Jie Y, Lin Y, Billot L, Munoz-Venturelli P, Martins S, Pontes-Neto OM, Liu L, Chalmers J, Carcel C, Song L, Anderson CS; INTERACT Investigators. Effects of blood pressure lowering in relation to time in acute intracerebral haemorrhage: a pooled analysis of the four INTERACT trials. Lancet Neurol. 2025 Jul;24(7):571-579. doi: 10.1016/S1474-4422(25)00160-7. PMID 40541207
- [Derived] Maegele M. Towards optimization in the use of hemostatic agents and blood products in the early treatment of patients with traumatic brain injury (TBI). Curr Opin Anaesthesiol. 2025 Apr 1;38(2):129-135. doi: 10.1097/ACO.0000000000001465. Epub 2025 Feb 14. PMID 39945652
- [Derived] You S, Zheng D, Yoshimura S, Ouyang M, Han Q, Wang X, Cao Y, Delcourt C, Song L, Arima H, Chen X, Liu CF, Lindley RI, Robinson T, Anderson CS, Chalmers J; INTERACT Investigators. Optimum Baseline Clinical Severity Scale Cut Points for Prognosticating Intracerebral Hemorrhage: INTERACT Studies. Stroke. 2024 Jan;55(1):139-145. doi: 10.1161/STROKEAHA.123.044538. Epub 2023 Nov 29. PMID 38018833
- [Derived] Sandset EC, Wang X, Carcel C, Sato S, Delcourt C, Arima H, Stapf C, Robinson T, Lavados P, Chalmers J, Woodward M, Anderson CS. Sex differences in treatment, radiological features and outcome after intracerebral haemorrhage: Pooled analysis of Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage trials 1 and 2. Eur Stroke J. 2020 Dec;5(4):345-350. doi: 10.1177/2396987320957513. Epub 2020 Sep 20. PMID 33598552
- [Derived] Wang X, Moullaali TJ, Li Q, Berge E, Robinson TG, Lindley R, Zheng D, Delcourt C, Arima H, Song L, Chen X, Yang J, Chalmers J, Anderson CS, Sandset EC. Utility-Weighted Modified Rankin Scale Scores for the Assessment of Stroke Outcome: Pooled Analysis of 20 000+ Patients. Stroke. 2020 Aug;51(8):2411-2417. doi: 10.1161/STROKEAHA.119.028523. Epub 2020 Jul 9. PMID 32640944
- [Derived] Wang X, Sandset EC, Moullaali TJ, Chen G, Song L, Carcel C, Delcourt C, Woodward M, Robinson T, Chalmers J, Arima H, Anderson CS; INTERACT2 Investigators. Determinants of the high admission blood pressure in mild-to-moderate acute intracerebral hemorrhage. J Hypertens. 2019 Jul;37(7):1463-1466. doi: 10.1097/HJH.0000000000002056. PMID 31085948
- [Derived] Chen R, Wang X, Anderson CS, Robinson T, Lavados PM, Lindley RI, Chalmers J, Delcourt C. Infratentorial Intracerebral Hemorrhage. Stroke. 2019 May;50(5):1257-1259. doi: 10.1161/STROKEAHA.118.023766. PMID 30890109
- [Derived] Delcourt C, Zheng D, Chen X, Hackett M, Arima H, Hata J, Heeley E, Al-Shahi Salman R, Woodward M, Huang Y, Robinson T, Lavados PM, Lindley RI, Stapf C, Davies L, Chalmers J, Anderson CS, Sato S; INTERACT Investigators. Associations with health-related quality of life after intracerebral haemorrhage: pooled analysis of INTERACT studies. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):70-75. doi: 10.1136/jnnp-2016-314414. Epub 2016 Oct 21. PMID 27919055
- [Derived] Song L, Sandset EC, Arima H, Heeley E, Delcourt C, Chen G, Yang J, Wu G, Wang X, Lavados PM, Huang Y, Stapf C, Wang J, Robinson TG, Chalmers J, Lindley RI, Anderson CS; INTERACT2 Investigators. Early blood pressure lowering in patients with intracerebral haemorrhage and prior use of antithrombotic agents: pooled analysis of the INTERACT studies. J Neurol Neurosurg Psychiatry. 2016 Dec;87(12):1330-1335. doi: 10.1136/jnnp-2016-313246. Epub 2016 May 13. PMID 27178897
- [Derived] Qiu M, Sato S, Zheng D, Wang X, Carcel C, Hirakawa Y, Sandset EC, Delcourt C, Arima H, Wang J, Chalmers J, Anderson CS; INTERACT Investigators*. Admission Heart Rate Predicts Poor Outcomes in Acute Intracerebral Hemorrhage: The Intensive Blood Pressure Reduction in Acute Cerebral Hemorrhage Trial Studies. Stroke. 2016 Jun;47(6):1479-85. doi: 10.1161/STROKEAHA.115.012382. Epub 2016 May 10. PMID 27165954
- [Derived] Moullaali TJ, Sato S, Wang X, Rabinstein AA, Arima H, Carcel C, Chen G, Robinson T, Heeley E, Chan E, Delcourt C, Stapf C, Cordonnier C, Lindley RI, Chalmers J, Anderson CS; INTERACT Investigators. Prognostic significance of delayed intraventricular haemorrhage in the INTERACT studies. J Neurol Neurosurg Psychiatry. 2017 Jan;88(1):19-24. doi: 10.1136/jnnp-2015-311562. Epub 2016 Jan 8. PMID 26746184
- [Derived] Wang X, Arima H, Al-Shahi Salman R, Woodward M, Heeley E, Stapf C, Lavados PM, Robinson T, Huang Y, Wang J, Delcourt C, Anderson CS. Rapid Blood Pressure Lowering According to Recovery at Different Time Intervals after Acute Intracerebral Hemorrhage: Pooled Analysis of the INTERACT Studies. Cerebrovasc Dis. 2015;39(3-4):242-8. doi: 10.1159/000381107. Epub 2015 Mar 25. PMID 25823544
- [Derived] Yang J, Arima H, Wu G, Heeley E, Delcourt C, Zhou J, Chen G, Wang X, Zhang S, Yu S, Chalmers J, Anderson CS; INTERACT Investigators. Prognostic significance of perihematomal edema in acute intracerebral hemorrhage: pooled analysis from the intensive blood pressure reduction in acute cerebral hemorrhage trial studies. Stroke. 2015 Apr;46(4):1009-13. doi: 10.1161/STROKEAHA.114.007154. Epub 2015 Feb 24. PMID 25712944
- [Derived] Priglinger M, Arima H, Anderson C, Krause M; INTERACT Investigators. No relationship of lipid-lowering agents to hematoma growth: pooled analysis of the intensive blood pressure reduction in acute cerebral hemorrhage trials studies. Stroke. 2015 Mar;46(3):857-9. doi: 10.1161/STROKEAHA.114.007664. Epub 2015 Feb 5. PMID 25657175
- [Derived] Sato S, Heeley E, Arima H, Delcourt C, Hirakawa Y, Pamidimukkala V, Li Z, Tao Q, Xu Y, Hennerici MG, Robinson T, Tzourio C, Lindley RI, Chalmers J, Anderson CS; INTERACT Investigators; Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang LJ, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J. Higher mortality in patients with right hemispheric intracerebral haemorrhage: INTERACT1 and 2. J Neurol Neurosurg Psychiatry. 2015 Dec;86(12):1319-23. doi: 10.1136/jnnp-2014-309870. Epub 2015 Jan 14. PMID 25589782
- [Derived] Wang X, Arima H, Al-Shahi Salman R, Woodward M, Heeley E, Stapf C, Lavados PM, Robinson T, Huang Y, Wang J, Delcourt C, Anderson CS; INTERACT Investigators. Clinical prediction algorithm (BRAIN) to determine risk of hematoma growth in acute intracerebral hemorrhage. Stroke. 2015 Feb;46(2):376-81. doi: 10.1161/STROKEAHA.114.006910. Epub 2014 Dec 11. PMID 25503550
- [Derived] Delcourt C, Huang Y, Arima H, Chalmers J, Davis SM, Heeley EL, Wang J, Parsons MW, Liu G, Anderson CS; INTERACT1 Investigators. Hematoma growth and outcomes in intracerebral hemorrhage: the INTERACT1 study. Neurology. 2012 Jul 24;79(4):314-9. doi: 10.1212/WNL.0b013e318260cbba. Epub 2012 Jun 27. PMID 22744655
- [Derived] Arima H, Huang Y, Wang JG, Heeley E, Delcourt C, Parsons M, Li Q, Neal B, Chalmers J, Anderson C; INTERACT1 Investigators. Earlier blood pressure-lowering and greater attenuation of hematoma growth in acute intracerebral hemorrhage: INTERACT pilot phase. Stroke. 2012 Aug;43(8):2236-8. doi: 10.1161/STROKEAHA.112.651422. Epub 2012 Jun 7. PMID 22678090
- [Derived] Arima H, Anderson CS, Wang JG, Huang Y, Heeley E, Neal B, Woodward M, Skulina C, Parsons MW, Peng B, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Morgenstern LB, Chalmers J; Intensive Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial Investigators. Lower treatment blood pressure is associated with greatest reduction in hematoma growth after acute intracerebral hemorrhage. Hypertension. 2010 Nov;56(5):852-8. doi: 10.1161/HYPERTENSIONAHA.110.154328. Epub 2010 Sep 7. PMID 20823381